CLINICAL TRIAL: NCT00182611
Title: Phase III Clinical Study of Preoperative S-1/CDDP Combination Chemotherapy in Patients With Potentially Resectable Stage III Advanced Gastric Cancer
Brief Title: S-1 and Cisplatin in Treating Patients Who Are Undergoing Surgery for Stage III Stomach Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyoto University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: KYUH-UHA-GC04-03; CDR0000426403 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2008-11

CONDITIONS: Gastric Cancer
Keywords: stage III gastric cancer; adenocarcinoma of the stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cisplatin; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Drug: cisplatin
Drug: tegafur-gimeracil-oteracil potassium
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as S-1 and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Giving chemotherapy before surgery may shrink the tumor so that it can be removed. It is not yet known whether giving S-1 together with cisplatin before surgery is more effective than surgery followed by S-1 in treating stomach cancer.

PURPOSE: This randomized phase III trial is studying how well giving S-1 together with cisplatin before surgery works compared to surgery followed by S-1 in treating patients with stage III stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall survival of patients with potentially resectable stage III gastric cancer treated with neoadjuvant S-1 and cisplatin followed by gastrectomy and adjuvant S-1 vs no neoadjuvant chemotherapy before gastrectomy and adjuvant S-1.

Secondary

* Compare the progression-free survival of patients treated with these regimens.
* Compare the curative resection rates in patients treated with these regimens.
* Compare the safety of these regimens, in terms of postoperative complications, adverse events, and treatment- or surgery-related mortality rate, in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease stage (T3 vs T4) and ECOG performance status (0 vs 1). Patients are randomized to 1 of 2 treatment arms.

* Arm I (control): Patients undergo gastrectomy with D2+ lymph node dissection. Patients then receive adjuvant oral S-1.
* Arm II (neoadjuvant therapy): Patients receive neoadjuvant oral S-1 on days 1-21 and cisplatin IV over 2 hours on day 8. Treatment repeats every 35 days for 2 courses in the absence of disease progression. Patients then undergo surgery and receive adjuvant S-1 as in arm I.

PROJECTED ACCRUAL: A total of 100 patients (50 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed gastric adenocarcinoma, including type II or type III adenocarcinoma of the esophagogastric junction

  * Stage III disease

    * T3 or T4 and/or N2

      * No stage IV disease
  * Helical CT scan and laparoscopic staging required
* Potentially resectable disease

PATIENT CHARACTERISTICS:

Age

* 20 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 4,000/mm³, but < 12,000/mm³
* Granulocyte count ≥ 2,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL

Hepatic

* AST and ALT ≤ 2.5 times upper limit of normal
* Bilirubin ≤ 1.5 mg/dL

Renal

* Creatinine clearance ≥ 50 mL/min

Pulmonary

* Arterial oxygen pressure (PaO_2) ≥ 70 mm Hg on room air

Other

* Able to take oral medications

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for gastric cancer

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for gastric cancer

Surgery

* No prior surgery for gastric cancer

Other

* No other prior therapy for gastric cancer

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-04; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Progression-free survival (PFS)
Postoperative PFS
Surgical/pathological curative resection
Death related to treatment
Death related to operation
Postoperative complications
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Seiji Satoh, Study Chair — Kyoto University Hospital
Locations (6):
- Japan (6):
  - Fukui Red Cross Hospital, Fukui-shi, Fukui
  - Kyoto University Hospital, Kyoto, Kyoto
  - National Hospital Organization - Kyoto Medical Center, Kyoto, Kyoto
  - Yamato Municipal Hospital, Yamatotakada, Nara
  - Kitano Hospital, Osaka, Osaka
  - Shimane Prefectural Central Hospital, Izumo-shi, Shimane